CLINICAL TRIAL: NCT03922555
Title: Phase I Trial of ASTX727 in Recurrent/Progressive Non-enhancing IDH Mutant Gliomas
Brief Title: ASTX727 in Recurrent/Progressive Non-enhancing IDH Mutant Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Isabel Arrillaga-Romany, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-631
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Neurological Cancer
Keywords: Neurological Cancer
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASTX727 (Cedazuridine + Cytidine Antimetabolite Decitabine) (Experimental): -ASTX727 administered orally for 5 or 6 consecutive days every 28d cycle and will de-escalate to 4 consecutive days every 28 d cycle.
  Interventions: Drug: ASTX727
- Expansion Cohort (Experimental): * Oral ASTX727 will be administered daily for 4, 5 or 6 consecutive days
  * Surgical resection will take place 12 days (+/- 1 day) after initiation of treatment
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: ASTX727 — ASTX727 is made up of the 2 study drugs cedazuridine and decitabine. Cedazuridine is believed to work by slowing down how fast decitabine is broken down by the body. Decitabine is believed to work by blocking abnormal cells or cancer cells from growing.

SUMMARY:
this research study is evaluating the highest dose of ASTX727 that can be administered safely to recurrent/progressive non-enhancing IDH mutant gliomas patients.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved ASTX727 as a treatment for any disease.

ASTX727 is made up of the 2 study drugs cedazuridine and decitabine. Cedazuridine is believed to work by slowing down how fast decitabine is broken down by the body. Decitabine is believed to work by blocking abnormal cells or cancer cells from growing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age.
* Participants must have histologically or cytologically confirmed glioma, with documented IDH1 and/or IDH2 gene-mutation.
* Participants must have radiographic evidence of non-enhancing disease progression/recurrence per RANO criteria for low grade gliomas (LGG).
* Patients who have received prior treatment with chemotherapy, radiation, or a combination of both are eligible. Also, patients who have not received any prior treatment for their glioma are also eligible.
* Participants must be ≥12 weeks from completion of radiation.
* Participants must have a baseline brain MRI scan within 28 days prior to Day 1 of treatment.
* Participants must be on a stable or decreasing dose of glucocorticoids for 7 days prior to registration.
* Participants must have archived primary tumor biopsies or surgical specimens for additional exploratory translational studies. At least 100-micron length of FFPE tissue or a tissue block should be available for enrollment and for shipment to the Sponsor, or a laboratory designated by the Principal Investigator. If less material is available, participants could still be eligible after discussion with the Principal Investigator who will assess and confirm that there is sufficient material for key evaluations.
* Participants must be able to understand and willing to sign an informed consent. A legally authorized representative may consent on behalf of a participant who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or site's Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Participants must have KPS ≥ to 70
* Participants must have expected survival of ≥ 6 months.
* Participants must have adequate bone marrow function as evidenced by:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥1500/mcL;
  * Hemoglobin ≥10 g/dL
  * Platelets ≥100,000/mcL
* Participants must have adequate hepatic function as evidenced by:

  * Serum total bilirubin ≤1.5 x upper limit of normal (ULN), unless considered due to Gilbert's disease
  * Aspartate aminotransferase (AST), Alanine Aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3.0 x ULN.
* Participants must have adequate renal function as evidenced by:

  * Serum creatinine ≤2.0 x ULN
  * OR Creatinine clearance >40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation: (140 - Age) × (weight in kg) × (0.85 if female)/72 × serum creatinine
* Participants must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer. (Participants with residual Grade 1 toxicity due to prior chemotherapy are allowed).
* Female participants with reproductive potential must have a negative serum pregnancy test within 14 days prior to the first study drug administration. Participants with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., have had menses at any time in the preceding 24 consecutive months). Women with reproductive potential as well as fertile men and their partners who are female with reproductive potential must agree to abstain from sexual intercourse or to use 2 effective forms of contraception from the time of giving informed consent, during the study, and for 90 days (females and males) following the last dose of ASTX727.
* Participants enrolling in the expansion cohort (Arm B) must meet all of the above criteria and must have surgically accessible tumors and be surgical candidates.

Exclusion Criteria:

* Participants with enhancing disease on brain MRI.
* Participants who received systemic anticancer therapy <28 days prior to registration. One exception: participants on lomustine/CCNU must wait at least 42 days from last date of drug administration to registration.
* Participants who received an investigational agent <14 days prior to registration. In addition, the first dose of ASTX727 should not occur before a period ≥5 half-lives of the investigational agent has elapsed.
* Participants with prior treatment with bevacizumab (Avastin) are excluded.
* Participants who are pregnant or breast-feeding.
* Participants with an active severe infection that requires anti-infective therapy or with an unexplained fever >38.5°C during screening visits or on their first day of study drug administration.
* Participants with known additional malignancy that is progressing or requires active treatment within 2 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer that has undergone potentially curative therapy, or surgically treated prostate cancer.
* Participants with known hypersensitivity to any of the components of ASTX727.
* Participants with a history of myocardial infarction within the 6 months prior to screening.
* Participants with a known history of severe and/or uncontrolled ventricular arrhythmias.
* Participants with QTc interval ≥450 msec or with other factors that significantly increase the risk of QT prolongation or arrhythmic events (e.g., family history of long QT interval syndrome).
* Participants with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C.
* Participants with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a participant's ability to sign informed consent, cooperate, or participate in the study.
* Participants with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Participants with evidence of intracranial or intratumoral hemorrhage either by MRI or CT scan. Participants with resolving post-surgical changes, punctate/micro-hemorrhage, or hemosiderin are eligible.
* Participants enrolling in the expansion cohort will be excluded is they are deemed by the treating physician or surgeon not to be suitable for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  Participants will be enrolled at escalating doses using a standard 3+3 dose escalation design until the maximum administered dose is reached or until dose limiting toxicities result in the end of dose escalation. The maximum tolerated dose is the highest administered dose level at which participants experienced experienced 1 or fewer dose limiting toxicities.

SECONDARY OUTCOMES:
Median Progression Free Survival | From the time of randomization until disease progression or death, up to five years
  Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Disease progression will be assessed using the Response Assessment in Neuro-Oncology (RANO) Working Group updated response assessment criteria for low-grade Gliomas.
Overall Survival | From the time of randomization until death, up to five years
  Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Response Rate | 1 Year
  The number of participants achieving a complete or partial tumor response as assessed using the the Response Assessment in Neuro-Oncology (RANO) Working Group updated response assessment criteria for low-grade Gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Arrillaga-Romany, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Dr. Isabel Arrillaga-Romany. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation